CLINICAL TRIAL: NCT01888146
Title: Collaborative Care for Chronic Pain in Primary Care
Brief Title: Pain Program for Active Coping & Training
Acronym: PPACT-UH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1UH2AT007788-01 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2013-06-27 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Non-malignant Pain
Keywords: Pain management; Opioid use; Pragmatic; Collaborative care; Primary care
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interdisciplinary pain program (Experimental): Interdisciplinary pain program, which includes behavioral health, nurse case management, physical therapy, and pharmacy embedded in primary care.
  Interventions: Behavioral: Interdisciplinary pain program
- Treatment as usual (No Intervention): Patients in this arm will receive care as usual and utilize services as they currently exist in the health plan system.

INTERVENTIONS:
Behavioral: Interdisciplinary pain program — Interdisciplinary pain program, which includes behavioral health, nurse case management, physical therapy, and pharmacy embedded in primary care.
  Arms: Interdisciplinary pain program

SUMMARY:
The overall aim of this study is to adopt an integrative rehabilitation approach for helping patients adopt self-management skills for managing chronic pain, limiting use of opioid medications, and identifying exacerbating factors amenable to treatment (e.g., depression, sleep problems) that is feasible and sustainable within the primary care setting.

DETAILED DESCRIPTION:
Pain is a common and very costly public health problem. Common chronic pain conditions are expensive and pervasive, affecting at least 116 million American adults at an annual cost of $560 billion in direct medical treatment costs and lost productivity, and disproportionally affect vulnerable populations. Pain is the primary reason patients seek medical care and, as the first point of contact, primary care providers (PCPs) deliver the majority of that care. Unfortunately, PCPs face many challenges in managing these patients' care and often have little specific training in pain medicine. Yet with proper system support, PCPs are in the best position to coordinate pain management longitudinally. While pharmacotherapy is the predominant treatment approach for many PCPs, this limits the patient's role to taking medication, and he or she can become a passive recipient of care-leading to poor outcomes, potential overmedication, and possible disillusionment with the medical system. Further, increases in opiate prescribing for pain treatment -amidst increasing awareness of adverse outcomes, including addiction-and limited efficacy suggest the importance of broader treatment approaches that focus on patients' improvement of functioning. Although opiates may reduce pain symptoms while prescribed, patients are unlikely to experience significant and sustained improvements without the use of other nonpharmacologic pain management approaches. Medical management of patients with persistent pain and complex problems is often fragmented, which leads patients to seek a wide variety of primary and specialty care services in an effort to manage their pain and related conditions. Such fragmented care leads to poorer outcomes and significantly increases health care costs as patients often receive unneeded diagnostic and medical procedures. While research has identified evidence-based multidisciplinary behavioral treatment approaches that are effective for such patients and can even prevent the disability associated with persistent pain when offered earlier in the course of care, these interventions are rarely available in everyday practice settings and will require data from pragmatic clinical trials to change the care paradigm.

To address these issues, we are proposing a mixed-methods, cluster-randomized pragmatic clinical trial that will evaluate the integration of psychosocial services within the primary care environment. This project will implement an intervention into everyday clinical practice flow utilizing assessment measures and intervention staff directly from the clinical care system rather than utilizing a research-developed and administered structure. The intervention will be an integrated program that will guide all care for intervention patients. We will compare this primary care-based intervention to usual care using systematic, clinic-based assessments. During the initial phase, we will pilot the intervention with up to 50 patients in the Kaiser Permanente Northwest (KPNW) region with patients selected by their primary care providers who have non-malignant chronic pain (pain persisting for ≥ 3 months) and who are on long-term opiate therapy for the treatment of their condition. This pilot portion of the project is in preparation for the effective implementation of a large-scale, cluster-randomized pragmatic clinical trial to be conducted throughout three regions of Kaiser Permanente - Northwest, Georgia, and Hawaii comparing this primary care based multidisciplinary intervention to usual care in these settings.

This intervention brings together elements often available in health plans but organized in a less integrated fashion, and it will ensure flexibility in implementation to best fit individual clinic environments and the needs of chronic pain patients on long-term opiate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Paneled to a primary care provider practicing at one of the primary care clinics participating in the study
* ≥18 years of age at time of inclusion. Current adult KP member (18 years or older)
* Within the last 180 days either:

  * 90 day supply of short acting opioid spanning at least 120 days
  * or more long acting opioid dispenses
* Pain diagnostic ICD-9 code within the past 180 days

  * Diagnostic categories include but are not limited to: Back pain, neck pain, fibromyalgia, arthritis, myofascial pain, neuropathies, migraine, tension headache, temporomandibular joint disorder, carpal tunnel syndrome, nonspecific chronic pain, abdominal pain, pelvic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Collected every 3 months for 1 year
  Reliable and valid tool that measures patients' pain intensity and functional interference.

SECONDARY OUTCOMES:
Health care utilization and cost | Collected every 3 months for 1 year
  Primary care and specialty care services

OTHER OUTCOMES:
Morphine equivalents | Collected every 3 months for 1 year
  Opioid dose measured in morphine equivalents
Patient satisfaction | Collected every 3 months for 1 year
  Patient satisfaction with health care services

CONTACTS AND LOCATIONS:
Overall Officials: Lynn DeBar, PhD, MHP, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States